CLINICAL TRIAL: NCT03104660
Title: Coronary and Structural Interventions Ulm - Transcatheter Mitral Valve Repair (CSI-Ulm-TMVR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Wohrle, Principal Investigator, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI-Ulm-TMVR
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: CE certified mitral valve repair systems
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CE certified mitral valve repair systems (Experimental): CE certified transcatheter mitral valve repair systems
  Interventions: Device: CE certified mitral valve repair systems

INTERVENTIONS:
Device: CE certified mitral valve repair systems — Patients receive a transcatheter mitral valve repair with CE certified transcatheter mitral repair systems.

SUMMARY:
To evaluate the long-term results after transcatheter mitral valve repair

DETAILED DESCRIPTION:
Patients with transcatheter mitral valve repair are followed for 10 years to demonstrate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* mitral valve regurgitation
* transcatheter mitral valve repair

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cerebral and cardiac events | 10 years
  Major adverse cerebral and cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Woehrle, MD, Principal Investigator — University Hospital Ulm
Locations (1):
- University Hospital Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seeger J, Markovic S, Kessler M, Rottbauer W, Wohrle J. Apixaban After Percutaneous Edge-to-Edge Mitral Valve Repair in Patients With Maintained Sinus Rhythm. JACC Cardiovasc Interv. 2019 Jan 28;12(2):214-216. doi: 10.1016/j.jcin.2018.11.009. No abstract available. PMID 30678801
- [Result] Seeger J, Muller P, Gonska B, Scharnbeck D, Markovic S, Walcher D, Rottbauer W, Wohrle J. Percutaneous Mitral Valve Repair With the MitraClip in Primary Compared With Secondary Mitral Valve Regurgitation Using the Mitral Valve Academic Research Consortium Criteria. J Invasive Cardiol. 2017 Apr;29(4):145-150. PMID 28368846